CLINICAL TRIAL: NCT03657147
Title: Improving African American Glaucoma Patient Involvement in Visits and Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 17-0688; 1R01HS025370-01 (AHRQ)
Record Dates: First submitted 2018-08-28; First posted 2018-09-04 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Question Prompt List and Video (Experimental): Participants will watch an educational video and question prompt list will be provided. Glaucoma visits will be audio-taped. A 15-20-minute interview will be conducted after the visit by a research assistant.
  Interventions: Behavioral: Educational Video and Question Prompt List
- Usual Care (No Intervention): The usual care group will not receive any intervention. Glaucoma visits will be audio-taped. A 15-20-minute interview will be conducted after the visit by a research assistant.

INTERVENTIONS:
Behavioral: Educational Video and Question Prompt List — A short educational video will be presented on an iPad about the importance of encouraging patients to ask questions and to be involved during glaucoma visits to improve self-management skills. A question prompt list will also be completed where participants check questions of interest to ask the provider.
  Arms: Question Prompt List and Video

SUMMARY:
This is a research project about services provided to African American patients with glaucoma. The goal of the project is to improve communication between providers and African-American patients about glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Age 18 or older
* Able to speak and read English
* Mentally competent to participate
* Not blind (are at least 20/400 in their better seeing eye)
* On one or more glaucoma medications
* Report being less than 80% adherent to their glaucoma medications on a Visual Analog Scale

Exclusion Criteria:

* < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure | 12 months
  Intraocular pressure measurements will be extracted from each patient's medical record at the baseline, 6 month, and 12 month follow-up visits. For all time points, a mean intraocular pressure will be calculated by averaging the intraocular pressure across both eyes. Change in intraocular pressure over the 12 month period will then be assessed by calculating the difference in mean intraocular pressure.
Glaucoma Medication Percent Adherence | 12 months
  Medication adherence will be measured using the number of recorded doses from the Medication Event Monitoring System (MEMS) data, divided by the number of prescribed doses. Medication adherence can range from 0% to 100%.
Glaucoma Medication Adherence Self-Efficacy Score | 12 months
  Medication adherence self-efficacy is measured using a 21-item scale that has a reliability of 0.89. Scores can range from 21 to 63, and a higher score indicates a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Betsy Sleath, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sleath B, Carpenter DM, Davis SA, Budenz DL, Muir KW, Romero MS, Lee C, Tudor G, Garcia N, Adjei AA, Robin AL. Improving Black Patient Question-Asking and Provider Education During Glaucoma Visits. Ophthalmol Glaucoma. 2023 Mar-Apr;6(2):206-214. doi: 10.1016/j.ogla.2022.09.003. Epub 2022 Sep 19. PMID 36967704
- [Derived] Sleath B, Carpenter DM, Budenz DL, Muir KW, Romero MS, Tudor G, Garcia N, Adjei AA, Robin AL. Provider use of a participatory decision-making style with African American patients with glaucoma. Patient Educ Couns. 2023 Jun;111:107679. doi: 10.1016/j.pec.2023.107679. Epub 2023 Feb 20. PMID 36848727
- [Derived] Sleath B, Carpenter DM, Davis SA, Budenz DL, Muir KW, Romero MS, Lee C, Tudor G, Garcia N, Adjei AA, Robin AL. Acceptance of a Pre-visit Intervention to Engage African American Glaucoma Patients during Visits. Optom Vis Sci. 2022 Dec 1;99(12):838-843. doi: 10.1097/OPX.0000000000001959. Epub 2022 Nov 26. PMID 36594752

DOCUMENTS (1):
  • Informed Consent Form (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT03657147/ICF_000.pdf